CLINICAL TRIAL: NCT03349580
Title: Early Initiation of a Strength Training Based Rehabilitation After Lumbar Spine Fusion Improves Core Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dejan Kernc (Other)
Collaborators: University Medical Centre Ljubljana (Other); University of Ljubljana (Other); Slovenian Research Agency (Other)
Responsible Party: Sponsor-Investigator, Dejan Kernc, Principal Investigator, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EarlyRehab-LSF
Record Dates: First submitted 2017-11-12; First posted 2017-11-21 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Lumbar Spine Fusion
Keywords: rehabilitation; randomized controlled trial; strength training; early initiation; intra-abdominal pressure

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The training group (Experimental): The training group performed rehabilitation program twice per week over 9 weeks. The group commenced rehabilitation 3 weeks after the surgery. During the phase one training (week 1 to week 5), the isometric exercises were preformed on the trunk extension, flexion and lateral flexion muscles. During the phase 2 (week 6 to week 9), the exercises were performed on the strength machines and duration of the exercises were maintained and prolonged to 30 seconds. The leg adduction and hip extension exercises were added. The patients were instructed to perform abdominal bracing (IAP) and maintain the neutral position of their lumbar spine before and during the exercises.
  Interventions: Behavioral: The training group
- The control group (No Intervention): The control group followed the hospital's standard protocol. These do not include exercises or physiotherapy before 3 months after surgery.

INTERVENTIONS:
Behavioral: The training group — The training group performed rehabilitation program twice per week over 9 weeks. The group commenced rehabilitation 3 weeks after the surgery. During the phase one training (week 1 to week 5), the isometric exercises were preformed on the trunk extension, flexion and lateral flexion muscles. During the phase 2 (week 6 to week 9), the exercises were performed on the strength machines and duration of the exercises were maintained and prolonged to 30 seconds. The leg adduction and hip extension exercises were added. The patients were instructed to perform abdominal bracing (IAP) and maintain the neutral position of their lumbar spine before and during the exercises.
  Arms: The training group

SUMMARY:
To analyze safety and the effects of early initiation of the rehabilitation. Including the objective measurement outcomes after lumbar spine fusion, based on the principles of strength training.

DETAILED DESCRIPTION:
The 27 patients were recruited for the study, aged 45 to 70 years, who had undergone lumbar spine fusion. The patients were randomized in to two groups. The strength training group started rehabilitation 3 weeks after surgery. The patients exercised two times per week, over 9 weeks. The focus was on muscle activation of lumbopelvic muscles stabilization. The control group followed a standard postoperative protocol, where no exercises were performed at the rehabilitation stage. The functional outcomes and the plain radiographs were evaluated after 3 weeks and subsequently after 3 and 18 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of degenerative, low-grade isthmic spondylolisthesis or degenerative disc disease with or without spinal stenosis.

Exclusion Criteria:

* Previous lumbar fusion surgery, degenerative or idiopathic scoliosis, inflammatory disease, and history of malignancy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change of isometric trunk muscle strength | Baseline, 9 weeks and 18 months.
  The isometric trunk muscle extension, flexion and lateral flexion strength were measured using a strain-gauge dynamometer. Maximum torque was calculated from the force sensor data (Newton) and the lever as a distance between the middle line of the belt and the iliac crest level (meter). A higher values represent a better outcome. The scale range were 48 Nm -830 Nm for extension, 12 Nm - 1010 Nm for flexion, 35 Nm - 680 Nm for lateral flexion right and 16 Nm - 640 Nm for lateral flexion left.
Change of low back pain disability as measured by the Oswestry Disability Index | Baseline, 9 weeks and 18 months.
  Self-reported levels of low back pain disability. The Oswestry Disability Index is presented as a score from 0 to 100 where lower scores represent lower levels of low back pain disability.

SECONDARY OUTCOMES:
Change of walking distance as measured by the 6-min walking test | Baseline, 9 weeks and 18 months.
  The walked distance was measured. A higher values represent a better outcome. The scale range was from 40m to 800m.
Change the repetition of stand-ups during the Chair stand test. | Baseline, 9 weeks and 18 months.
  A number of stand-ups in 30 seconds. A higher values represent a better outcome. The scale range was from 1 to 29 repetitions.
Change of height as measured by the Standing reach height test. | Baseline, 9 weeks and 18 months.
  A height which someone can reach. A higher values represent a better outcome. The scale range was from 190cm to 236cm.
Change of Intra-abdominal pressure pre-activation pattern. | Baseline, 9 weeks and 18 months.
  A lateral abdominal force sensor was used to estimate the time delay between the start of the increase in intra-abdominal pressure and the start of the force rise from the force plate (action start). The initiation of intra-abdominal pressure before starting the action contributed to better performance and result. The scale range was from -0.7s to 0.7s.
Change of pain disability as measured by the Visual Analogue Scale. | Baseline, 9 weeks and 18 months.
  Self-reported levels of pain disability. The Visual Analogue Scale presents back pain intensity with scores from 0 to 10, where 0 = "no problems" and 10 = "maximum problems".

CONTACTS AND LOCATIONS:
Overall Officials: Rok Vengust, Phd, Study Chair — University Medical Centre Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christensen FB, Laurberg I, Bunger CE. Importance of the back-cafe concept to rehabilitation after lumbar spinal fusion: a randomized clinical study with a 2-year follow-up. Spine (Phila Pa 1976). 2003 Dec 1;28(23):2561-9. doi: 10.1097/01.BRS.0000097890.96524.A1. PMID 14652472
- [Background] Nielsen PR, Jorgensen LD, Dahl B, Pedersen T, Tonnesen H. Prehabilitation and early rehabilitation after spinal surgery: randomized clinical trial. Clin Rehabil. 2010 Feb;24(2):137-48. doi: 10.1177/0269215509347432. PMID 20103575
- [Background] Greenwood J, McGregor A, Jones F, Mullane J, Hurley M. Rehabilitation Following Lumbar Fusion Surgery: A Systematic Review and Meta-Analysis. Spine (Phila Pa 1976). 2016 Jan;41(1):E28-36. doi: 10.1097/BRS.0000000000001132. PMID 26555833
- [Background] Oestergaard LG, Nielsen CV, Bunger CE, Svidt K, Christensen FB. The effect of timing of rehabilitation on physical performance after lumbar spinal fusion: a randomized clinical study. Eur Spine J. 2013 Aug;22(8):1884-90. doi: 10.1007/s00586-013-2717-5. Epub 2013 Apr 6. PMID 23563500
- [Background] Oestergaard LG, Christensen FB, Nielsen CV, Bunger CE, Fruensgaard S, Sogaard R. Early versus late initiation of rehabilitation after lumbar spinal fusion: economic evaluation alongside a randomized controlled trial. Spine (Phila Pa 1976). 2013 Nov 1;38(23):1979-85. doi: 10.1097/BRS.0b013e3182a7902c. PMID 23928716
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Hanscom B, Tosteson AN, Blood EA, Birkmeyer NJ, Hilibrand AS, Herkowitz H, Cammisa FP, Albert TJ, Emery SE, Lenke LG, Abdu WA, Longley M, Errico TJ, Hu SS. Surgical versus nonsurgical treatment for lumbar degenerative spondylolisthesis. N Engl J Med. 2007 May 31;356(22):2257-70. doi: 10.1056/NEJMoa070302. PMID 17538085
- [Background] Deyo RA, Gray DT, Kreuter W, Mirza S, Martin BI. United States trends in lumbar fusion surgery for degenerative conditions. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1441-5; discussion 1446-7. doi: 10.1097/01.brs.0000166503.37969.8a. PMID 15959375
- [Background] Cholewicki J, Juluru K, McGill SM. Intra-abdominal pressure mechanism for stabilizing the lumbar spine. J Biomech. 1999 Jan;32(1):13-7. doi: 10.1016/s0021-9290(98)00129-8. PMID 10050947
- [Background] Hodges PW, Cresswell AG, Daggfeldt K, Thorstensson A. In vivo measurement of the effect of intra-abdominal pressure on the human spine. J Biomech. 2001 Mar;34(3):347-53. doi: 10.1016/s0021-9290(00)00206-2. PMID 11182126
- [Background] Oestergaard LG, Nielsen CV, Bunger CE, Sogaard R, Fruensgaard S, Helmig P, Christensen FB. The effect of early initiation of rehabilitation after lumbar spinal fusion: a randomized clinical study. Spine (Phila Pa 1976). 2012 Oct 1;37(21):1803-9. doi: 10.1097/BRS.0b013e31825a17ab. PMID 22565381
- [Background] Abbott AD, Tyni-Lenne R, Hedlund R. Early rehabilitation targeting cognition, behavior, and motor function after lumbar fusion: a randomized controlled trial. Spine (Phila Pa 1976). 2010 Apr 15;35(8):848-57. doi: 10.1097/BRS.0b013e3181d1049f. PMID 20354468
- [Derived] Kernc D, Strojnik V, Vengust R. Early initiation of a strength training based rehabilitation after lumbar spine fusion improves core muscle strength: a randomized controlled trial. J Orthop Surg Res. 2018 Jun 19;13(1):151. doi: 10.1186/s13018-018-0853-7. PMID 29914580